CLINICAL TRIAL: NCT01522053
Title: Comparison of the Catheter-over-needle and Catheter-through-needle Methods for Continuous Delivery of Local Anesthetic During Peripheral Nerve Blockade
Brief Title: Catheter-over-needle: Inpatient Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI no longer at institution
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro000027409
Record Dates: First submitted 2012-01-26; First posted 2012-01-31 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Local Anesthesia; Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Catheter-over-needle (Experimental): Patients will receive a catheter placed by a catheter-over-needle method.
  Interventions: Procedure: Catheter-over-needle
- Catheter-through-needle (Active Comparator): Patients will receive a catheter placed by the traditional catheter-though-needle method.
  Interventions: Procedure: Catheter-through-needle

INTERVENTIONS:
Procedure: Catheter-over-needle — Patients in the experimental group will receive a perineural catheter placed by the catheter-over-needle method.
  Arms: Catheter-over-needle
Procedure: Catheter-through-needle — Patients in the control group will receive a perineural catheter placed by the traditional catheter-though-needle method.
  Arms: Catheter-through-needle

SUMMARY:
When anesthesiologists perform a regional nerve block, they will often put a catheter - a flexible plastic tube - in the patient to allow for continuous delivery of local anesthetic. This allows the nerve(s) to be 'frozen' so that the patient is more comfortable during and after surgery. The most common method of placing the catheter close to a nerve involves threading the catheter through a needle which has been inserted under the skin. Because the catheter is very thin and flexible, it does not thread well through tissue and will buckle and kink when enough force is applied to it. Another problem is that the puncture hole left by the needle is larger than the diameter of the catheter, meaning that when the needle is withdrawn, the catheter is not secure, which increases the chance that it will dislodge and cause leakage of local anesthetic. One solution to these problems is to use a catheter placement method similar to how intravenous catheters are installed. In this method, the catheter fits around ('over') the needle, which results in more support for the catheter while it is being pushed under the skin. We wish to examine if a catheter-over-needle method would be useful for placing a catheter to deliver local anesthetic during peripheral nerve blockade. We will compare the catheter-over-needle method to the currently used catheter-through-needle method on patients who require continuous anesthetic delivery for their surgery; half the patients will receive anesthetic through one method, and the other half will receive anesthetic through the other method. We believe that using the catheter-over-needle method will result in more secure placement of the catheter and more efficient delivery of local anesthetic.

DETAILED DESCRIPTION:
Background: Current needle-catheter assemblies are designed so that a flexible catheter is threaded through a larger diameter needle towards a target nerve. These catheter-through-needle (CTN) assemblies suffer from several fundamental problems, including leakage at the insertion site and dislodgement of the catheter. The underlying problem of this design is that the needle puncture hole is wider in diameter than the catheter diameter. An alternative catheter-over-needle (CON) design, in which the catheter diameter is larger than that of the needle puncture hole, may be a potential solution to the problems of leakage and dislodgement. We wish to evaluate the ease of use and effectiveness of the CON method in the clinical setting by having anesthesiologists perform and rate the two techniques during and after administration of local anesthesia at various block sites on the body.

Study objective: To compare the ease of use and effectiveness of the CON technique to the CTN method in delivering continuous local anesthesia during regional nerve blockade.

Hypothesis: Insertion of a CON assembly catheter will result in more secure and accurate catheter placement and more efficient delivery of local anesthetic compared to a catheter placed using the CTN method.

Primary outcomes:

1. Time taken to place catheter near target nerve after initial skin puncture.
2. Confidence in accurate catheter placement.
3. Assessment of catheter stability at insertion site.
4. Incidence of anesthetic/fluid leakage at catheter insertion site.

Study procedures: This study will involve recruiting patients who are scheduled to undergo surgery that requires a regional nerve block via local anesthetic delivery through a perineural catheter. We wish to compare the CON and CTN catheterization methods for delivering local anesthetic during common regional blocks. One hundred patients will be recruited to assess the usefulness of the CON method in delivering local anesthetic. Patients in the study group will receive a continuous infusion of local anesthetic through a CON catheter. Patients in the control group will receive continuous local anesthetic through a CTN catheter. To make data collection easier, we will perform assessments at several locations in the Edmonton zone; anesthesiologists at each location will be asked to participate in performing the blocks and record their assessment of the two catheterization methods.

On the day of surgery, patients will be taken to the regional block area, where they will be positioned appropriately for the block they are to receive. Under ultrasound guidance, the attending anesthesiologist will install either the CON or CTN catheter. Each CTN catheter will be inserted as per standard procedures; CON catheters will be inserted in a similar fashion to that used for intravenous catheters. The anesthesiologist will be given Part 1 of a survey to evaluate the catheterization technique. On this survey, they will record the duration of time from initial skin puncture to placement of the end of the catheter near the target nerve and provide a subjective evaluation of how confident they are in the accuracy of the catheter's placement. Following connection of a continuous infusion of local anesthetic, the anesthesiologist will record an assessment of catheter stability and incidence of anesthetic leakage around the catheter insertion site.

During the postoperative period, the anesthesiologist will complete Part 2 of the assessment survey, which will record their personal opinion on the CON method's ease of use and its value in the clinical setting.

Inclusion criteria: Adult; scheduled for surgery that requires peripheral nerve blockade

Exclusion criteria: Failure to provide informed consent; allergy to local anesthetic; neurological pathology and/or deficit in the block region.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 yrs)
* Scheduled for surgery that requires continuous peripheral nerve block

Exclusion Criteria:

* Failure to provide informed consent
* Allergy to local anesthetic
* Neurological pathology and/or deficit in the block region

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Incidence of anesthetic/fluid leakage at catheter insertion site. | Duration of time that perineural catheter is in the patient
  Evidence of leakage of local anesthetic at the catheter insertion site and any catheter dislodgement or premature withdrawal will be recorded.

SECONDARY OUTCOMES:
Confidence in accurate catheter placement. | Duration of catheter placement in patient.
  A subjective assessment of the catheterization and local anesthetic delivery technique will be provided by the anesthesiologist.
Time taken to place catheter near target nerve after initial skin puncture. | From identification of needle insertion site to correct placement of needle in patient; approximately 2 minutes.
  The time (in seconds) taken to correctly place the needle/catheter for delivery of local anesthetic will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Ip VH, Rockley MC, Tsui BC. The catheter-over-needle assembly offers greater stability and less leakage compared with the traditional counterpart in continuous interscalene nerve blocks: a randomized patient-blinded study. Can J Anaesth. 2013 Dec;60(12):1272-3. doi: 10.1007/s12630-013-0032-6. Epub 2013 Sep 17. No abstract available. PMID 24043379